CLINICAL TRIAL: NCT00947310
Title: IDE-Exempt: Multicenter Automatic Defibrillator Implantation Trial - Reduce Inappropriate Therapy
Brief Title: Multicenter Automatic Defibrillator Implantation Trial - Reduce Inappropriate Therapy
Acronym: MADIT-RIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MADIT-RIT
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2013-03

CONDITIONS: Primary Prevention of Sudden Cardiac Arrest
Keywords: Inappropriate therapy; ICD therapy; Primary prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Standard ICD Programming
  Interventions: Device: Standard ICD programming
- B (Experimental): High rate cutoff
  Interventions: Device: High rate cutoff
- C (Experimental): Long ICD duration delay
  Interventions: Device: Long delay

INTERVENTIONS:
Device: Standard ICD programming — Standard ICD programming
  Arms: A
Device: High rate cutoff — Programming of a high rate cutoff
  Arms: B
Device: Long delay — Programming of a prolonged delay
  Arms: C

SUMMARY:
This study will assess the impact of higher rate cutoffs and longer delays than standard programming on inappropriate therapy in primary prevention ICD and CRT-D patients.

DETAILED DESCRIPTION:
The purpose of the MADIT-RIT trial is to compare the time to first inappropriate therapy using high rate cutoff and/or long delay in primary prevention patients receiving an ICD or CRT-D device compared to standard programming.

ELIGIBILITY:
Inclusion Criteria:

* Primary prevention patient with ischemic or non-ischemic heart disease who meets current guidelines for dual-chamber ICD or CRT-D device therapy
* Patient in sinus rhythm
* Patient on stable optimal pharmacologic therapy for the cardiac condition or who has developed a recent ICD indication that necessitates ICD therapy concurrent with the optimization of pharmacologic therapy
* Patient ≥ 21 years of age, or legal representative, willing and capable of giving informed consent

Exclusion Criteria:

* Patient with an implanted pacemaker or CRT-P
* Patient with existing ICD or CRT-D device components
* Patient with a history of VT or VF
* Patient with permanent or chronic AF, or cardioversion for AF, within the past three calendar months before enrollment
* Patient with coronary artery bypass graft surgery or percutaneous coronary intervention within the past three calendar months prior to enrollment
* Patient with enzyme-positive myocardial infarction within the past three calendar months prior to enrollment
* Patient with angiographic evidence of coronary disease who are candidates for coronary revascularization and are likely to undergo coronary artery bypass graft surgery or percutaneous coronary intervention in the foreseeable future
* Patient with second or third degree heart block
* Patient in NYHA Class IV
* Patient who is pregnant or plans to become pregnant during the course of the trial
* Patient with irreversible brain damage from preexisting cerebral disease
* Patient with presence of any disease, other than the patient's cardiac disease, associated with a reduced likelihood of survival for the duration of the trial, e.g., cancer, uremia, liver failure, etc.
* Patient with chronic renal disease with BUN ≥ 50mg/dl or creatinine ≥ 2.5 mg/dl
* Patient participating in any other clinical trial
* Patient unwilling or unable to cooperate with the protocol
* Patient who lives at such a distance from the clinic that travel for follow-up visits would be unusually difficult
* Patient who does not anticipate being a resident of the area for the scheduled duration of the trial
* Patient unwilling to sign the consent for participation
* Patient whose physician does not allow participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Moss, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester (Multiple Facilities Participating World Wide), Rochester, New York, United States

REFERENCES:
- [Background] Schuger C, Daubert JP, Brown MW, Cannom D, Estes NA 3rd, Hall WJ, Kayser T, Klein H, Olshansky B, Power KA, Wilber D, Zareba W, Moss AJ. Multicenter automatic defibrillator implantation trial: reduce inappropriate therapy (MADIT-RIT): background, rationale, and clinical protocol. Ann Noninvasive Electrocardiol. 2012 Jul;17(3):176-85. doi: 10.1111/j.1542-474X.2012.00531.x. PMID 22816536
- [Derived] Younis A, Heist EK, McNitt S, Aktas MK, Rosero S, Goldenberg I, Kutyifa V. Predictors and outcomes of atrial tachyarrhythmia among patients with implantable defibrillators. Heart Rhythm. 2020 Apr;17(4):553-559. doi: 10.1016/j.hrthm.2019.11.024. Epub 2019 Nov 22. PMID 31765809
- [Derived] Jackson LR 2nd, Thomas KL, Polonsky B, Zareba W, Lahiri M, Saba S, McNitt S, Schuger C, Daubert JP, Moss AJ, Kutyifa V. Effectiveness of high rate and delayed detection ICD programming by race: A MADIT-RIT substudy. J Cardiovasc Electrophysiol. 2018 Oct;29(10):1418-1424. doi: 10.1111/jce.13693. Epub 2018 Jul 24. PMID 29978932
- [Derived] Kutyifa V, Daubert JP, Schuger C, Goldenberg I, Klein H, Aktas MK, McNitt S, Stockburger M, Merkely B, Zareba W, Moss AJ. Novel ICD Programming and Inappropriate ICD Therapy in CRT-D Versus ICD Patients: A MADIT-RIT Sub-Study. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e001965. doi: 10.1161/CIRCEP.114.001965. PMID 26743237
- [Derived] Kutyifa V, Daubert JP, Olshansky B, Huang DT, Zhang C, Ruwald AC, McNitt S, Zareba W, Moss AJ, Schuger C. Characterization and predictors of first and subsequent inappropriate ICD therapy by heart rate ranges: Result of the MADIT-RIT efficacy analysis. Heart Rhythm. 2015 Sep;12(9):2030-7. doi: 10.1016/j.hrthm.2015.05.021. Epub 2015 May 19. PMID 26001510
- [Derived] Kutyifa V, Moss AJ, Schuger C, McNitt S, Polonsky B, Ruwald AH, Ruwald MH, Daubert JP, Zareba W. Reduction in Inappropriate ICD Therapy in MADIT-RIT Patients Without History of Atrial Tachyarrhythmia. J Cardiovasc Electrophysiol. 2015 Aug;26(8):879-884. doi: 10.1111/jce.12692. Epub 2015 Jun 15. PMID 25917337
- [Derived] Stockburger M, Moss AJ, Olshansky B, Klein H, McNitt S, Schuger C, Daubert JP, Goldenberg I, Ruwald AC, Merkely B, Zareba W, Kutyifa V. Time-dependent risk reduction of ventricular tachyarrhythmias in cardiac resynchronization therapy patients: a MADIT-RIT sub-study. Europace. 2015 Jul;17(7):1085-91. doi: 10.1093/europace/euv008. Epub 2015 Mar 4. PMID 25745075
- [Derived] Sedlacek K, Ruwald AC, Kutyifa V, McNitt S, Thomsen PEB, Klein H, Stockburger M, Wichterle D, Merkely B, DE LA Concha JF, Swissa M, Zareba W, Moss AJ, Kautzner J, Ruwald MH; MADIT-RIT Investigators. The effect of ICD programming on inappropriate and appropriate ICD Therapies in ischemic and nonischemic cardiomyopathy: the MADIT-RIT trial. J Cardiovasc Electrophysiol. 2015 Apr;26(4):424-433. doi: 10.1111/jce.12605. Epub 2015 Feb 11. PMID 25546486
- [Derived] Ruwald AC, Schuger C, Moss AJ, Kutyifa V, Olshansky B, Greenberg H, Cannom DS, Estes NA, Ruwald MH, Huang DT, Klein H, McNitt S, Beck CA, Goldstein R, Brown MW, Kautzner J, Shoda M, Wilber D, Zareba W, Daubert JP. Mortality reduction in relation to implantable cardioverter defibrillator programming in the Multicenter Automatic Defibrillator Implantation Trial-Reduce Inappropriate Therapy (MADIT-RIT). Circ Arrhythm Electrophysiol. 2014 Oct;7(5):785-92. doi: 10.1161/CIRCEP.114.001623. Epub 2014 Aug 18. PMID 25136077
- [Derived] Ruwald MH, Okumura K, Kimura T, Aonuma K, Shoda M, Kutyifa V, Ruwald AC, McNitt S, Zareba W, Moss AJ. Syncope in high-risk cardiomyopathy patients with implantable defibrillators: frequency, risk factors, mechanisms, and association with mortality: results from the multicenter automatic defibrillator implantation trial-reduce inappropriate therapy (MADIT-RIT) study. Circulation. 2014 Feb 4;129(5):545-52. doi: 10.1161/CIRCULATIONAHA.113.004196. Epub 2013 Nov 7. PMID 24201303
- [Derived] Ruwald MH, Zareba W, Jons C, Zhang C, Ruwald AC, Olshansky B, McNitt S, Bloch Thomsen PE, Shoda M, Merkely B, Moss AJ, Kutyifa V. Influence of diabetes mellitus on inappropriate and appropriate implantable cardioverter-defibrillator therapy and mortality in the Multicenter Automatic Defibrillator Implantation Trial-Reduce Inappropriate Therapy (MADIT-RIT) Trial. Circulation. 2013 Aug 13;128(7):694-701. doi: 10.1161/CIRCULATIONAHA.113.002472. Epub 2013 Jul 23. PMID 23881862
- [Derived] Moss AJ, Schuger C, Beck CA, Brown MW, Cannom DS, Daubert JP, Estes NA 3rd, Greenberg H, Hall WJ, Huang DT, Kautzner J, Klein H, McNitt S, Olshansky B, Shoda M, Wilber D, Zareba W; MADIT-RIT Trial Investigators. Reduction in inappropriate therapy and mortality through ICD programming. N Engl J Med. 2012 Dec 13;367(24):2275-83. doi: 10.1056/NEJMoa1211107. Epub 2012 Nov 6. PMID 23131066

RESULTS

PARTICIPANT FLOW:
Groups:
- A - Standard ICD Programming: Standard ICD Programming
  Standard ICD programming : Standard ICD programming
- B - High Rate Cutoff: High rate cutoff
  High rate cutoff : Programming of a high rate cutoff
- C - Long ICD Duration Delay: Long ICD duration delay
  Long delay : Programming of a prolonged delay
Period: Overall Study
Arm/Group | A - Standard ICD Programming | B - High Rate Cutoff | C - Long ICD Duration Delay
Started | 514 | 500 | 486
Completed | 514 | 500 | 486
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Standard ICD Programming | B - High Rate Cutoff | C - Long ICD Duration Delay | Total
Number analyzed (Participants) | 514 | 500 | 486 | 1500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 252 | 245 | 254 | 751
  >=65 years | 262 | 255 | 232 | 749
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11) | 63 (12) | 62 (12) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 146 | 133 | 436
  Male | 357 | 354 | 353 | 1064
Region of Enrollment [Number; unit: participants]
  United States | 353 | 338 | 325 | 1016
  Europe | 94 | 92 | 91 | 277
  Japan | 22 | 22 | 24 | 68
  Canada | 11 | 12 | 12 | 35
  Israel | 34 | 36 | 34 | 104

OUTCOME MEASURES:

1. Secondary Outcome: All-cause Mortality
Time Frame: Average 1.4 years of follow-up
Measure: Number; unit: participants
Arm/Group | A - Standard ICD Programming | B - High Rate Cutoff | C - Long ICD Duration Delay
Number analyzed (Participants) | 514 | 500 | 486
participants | 34 | 16 | 21
Statistical Analysis 1: Comparison: A - Standard ICD Programming vs B - High Rate Cutoff; Hazard ratios (HR) were calculated to compare Arm A vs Arm B. Null Hypothesis was that HR = 1; Test type: Superiority or Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.24 to 0.85]
Statistical Analysis 2: Comparison: A - Standard ICD Programming vs C - Long ICD Duration Delay; Hazard ratios (HR) were calculated to compare Arm A vs Arm C. Null Hypothesis was that HR = 1; Test type: Superiority or Other; p = 0.06, Regression, Cox; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.30 to 1.02]

2. Secondary Outcome: Syncope
Description: First episode of syncope
Time Frame: Average of 1.4 years follow-up
Measure: Number; unit: participants
Arm/Group | A - Standard ICD Programming | B - High Rate Cutoff | C - Long ICD Duration Delay
Number analyzed (Participants) | 514 | 500 | 486
participants | 23 | 22 | 22
Statistical Analysis 1: Comparison: A - Standard ICD Programming vs B - High Rate Cutoff; Hazard ratios (HR) were calculated to compare Arm A vs Arm B. Null Hypothesis was that HR = 1; Test type: Superiority or Other; p = 0.39, Regression, Cox; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.71 to 2.47]
Statistical Analysis 2: Comparison: A - Standard ICD Programming vs C - Long ICD Duration Delay; Hazard ratios (HR) were calculated to compare Arm A vs Arm C. Null Hypothesis was that HR = 1; Test type: Superiority or Other; p = 0.80, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.58 to 2.05]

3. Primary Outcome: Inappropriate ICD Therapy
Description: First occurance of inappropriate therapy (either anti-tachycardia pacing or shock)
Time Frame: Average of 1.4 years follow-up
Measure: Number; unit: participants
Arm/Group | A - Standard ICD Programming | B - High Rate Cutoff | C - Long ICD Duration Delay
Number analyzed (Participants) | 514 | 500 | 486
participants | 105 | 21 [0.13 to 0.34] | 26 [0.15 to 0.40]
Statistical Analysis 1: Comparison: A - Standard ICD Programming vs B - High Rate Cutoff; Hazard ratios (HR) were calculated to compare Arm A vs Arm B. Null Hypothesis was that HR = 1; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.13 to 0.34]
Statistical Analysis 2: Comparison: A - Standard ICD Programming vs C - Long ICD Duration Delay; Hazard ratios (HR) were calculated to compare Arm A vs Arm C. Null Hypothesis was that HR = 1; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.15 to 0.40]

ADVERSE EVENTS:
Arm/Group | A - Standard ICD Programming | B - High Rate Cutoff | C - Long ICD Duration Delay
Serious Adverse Events (participants affected / at risk) | 446/514 | 380/500 | 394/486
Other Adverse Events (participants affected / at risk) | 207/514 | 136/500 | 121/486
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Standard ICD Programming (N=514) | B - High Rate Cutoff (N=500) | C - Long ICD Duration Delay (N=486)
Hematological (Blood and lymphatic system disorders) | 5 (7) | 3 (3) | 3 (3)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Thromboembolic events (Blood and lymphatic system disorders) | 18 (20) | 18 (18) | 15 (16)
Extracardiac Stimulation, Left Ventricular (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Lead Dislodgment, Left Ventricular (Cardiac disorders) | 11 (11) | 7 (7) | 11 (11)
Threshold Related, Left Ventricular (Cardiac disorders) | 5 (5) | 1 (1) | 3 (3)
Pulse Generator-System, Patient-Other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pacemaker-mediated Tachycardia (PMT) (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Unable to Communicate with Pulse Generator (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Threshold, Right Atrial (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Lead Dislodgment, Right Atrial (Cardiac disorders) | 7 (7) | 6 (6) | 5 (5)
Lead Related, Right Atrial (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Sensing Related, Right Atrial (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lead Dislodgment, Right Ventricular (Cardiac disorders) | 1 (1) | 9 (9) | 5 (7)
Lead Related, Right Ventricular (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Sensing Related, Right Ventricular (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Threshold Related, Right Ventricular (Cardiac disorders) | 3 (3) | 5 (5) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 4 (4) | 0 (0) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Chest Pain, Ischemic (Cardiac disorders) | 2 (2) | 6 (6) | 15 (17)
Chest Pain, Other (Cardiac disorders) | 12 (15) | 16 (17) | 17 (18)
Pulse Generator Erosion (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1)
Heart Failure Symptoms (Cardiac disorders) | 84 (141) | 67 (111) | 80 (130)
Hypertension (Cardiac disorders) | 2 (4) | 3 (3) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2) | 2 (3) | 6 (6)
Inappropriate Tachy Therapy (Cardiac disorders) | 14 (15) | 5 (5) | 2 (2)
Inadvertant Tachy Arrhythmia (Cardiac disorders) | 1 (1) | 4 (4) | 2 (2)
Pulse Generator Migration (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 7 (8) | 5 (6) | 5 (5)
Cardiovascular, Patient Condition (Cardiac disorders) | 12 (13) | 11 (13) | 8 (10)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Supraventricular Tachy Arrhythmia (Cardiac disorders) | 20 (25) | 17 (20) | 22 (29)
Valvular Related (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ventricular Arrhythmias (Cardiac disorders) | 26 (28) | 13 (15) | 15 (17)
Syncope, Cardiac Related (Cardiac disorders) | 4 (4) | 4 (5) | 4 (4)
Endocrine Related (Endocrine disorders) | 4 (4) | 3 (3) | 5 (8)
Gastrointestinal Related (Gastrointestinal disorders) | 28 (30) | 24 (33) | 25 (28)
Abnormal Laboratory Value (General disorders) | 5 (6) | 5 (5) | 5 (5)
Death (General disorders) | 1 (1) | 4 (4) | 4 (4) — This is not a complete listing of reported deaths, others are reported within other adverse event categories with a result in death.
Dizziness (General disorders) | 3 (3) | 4 (4) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (2) | 3 (3)
Head, Eyes, Ears, Nose, Throat (HEENT) (General disorders) | 4 (4) | 3 (3) | 6 (6)
Multi-System Failure (General disorders) | 1 (1) | 1 (1) | 3 (3)
Related to Multiple Symptoms (General disorders) | 5 (5) | 0 (0) | 2 (2)
Non-Cardiovascular, Patient Condition (General disorders) | 2 (2) | 6 (8) | 5 (5)
Physical Trauma (General disorders) | 7 (7) | 5 (5) | 8 (8)
Psychological (General disorders) | 3 (3) | 1 (1) | 0 (0)
Cancer (General disorders) | 6 (6) | 5 (5) | 7 (8)
Syncope, General (General disorders) | 3 (3) | 4 (4) | 2 (2)
Immune (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Systemic Infection (Infections and infestations) | 3 (3) | 6 (6) | 7 (7)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 15 (16) | 17 (17) | 10 (12)
Neurological (Nervous system disorders) | 8 (9) | 3 (3) | 5 (7)
Syncope, Neurological Related (Nervous system disorders) | 2 (2) | 1 (1) | 1 (2)
Genitourinary (Renal and urinary disorders) | 10 (12) | 7 (7) | 2 (3)
Renal (Renal and urinary disorders) | 14 (14) | 5 (5) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 7 (7) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 18 (22) | 20 (22) | 16 (16)
Integumentary (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (4) | 3 (3)
Myocardial Perforation, Post-Implant, Right Ventricular (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Seroma, Pocket (<= 30 days Post Pulse Generator Implant) (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Adverse Reaction, Implant Procedure Related (Surgical and medical procedures) | 2 (3) | 4 (5) | 0 (0)
Bleeding, Implant Procedure Related (Surgical and medical procedures) | 5 (5) | 2 (2) | 2 (2)
Coronary Venous Trauma (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hematoma, Pulse Generator Pocket (>30 days Post Device Implant) (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Infection, (> 30 days Post Device Implant) (Surgical and medical procedures) | 6 (6) | 5 (5) | 4 (4)
Pneumothorax, Procedure Related (Surgical and medical procedures) | 5 (5) | 5 (5) | 1 (1)
Post Surgical Wound Discomfort (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1)
Post Surgical Infection (<= 30 days Post Device Implant) (Surgical and medical procedures) | 3 (3) | 4 (4) | 3 (3)
Post Surgical Pocket Hemorrhage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Venous Occlusion (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Vascular Related (Vascular disorders) | 7 (10) | 4 (4) | 10 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Standard ICD Programming (N=514) | B - High Rate Cutoff (N=500) | C - Long ICD Duration Delay (N=486)
Extracardiac Stimulation, Left Ventricular (Cardiac disorders) | 32 (38) | 26 (28) | 24 (25)
Heart Failure Symptoms (Cardiac disorders) | 34 (44) | 32 (37) | 35 (39)
Inappropriate Tachy Therapy (Cardiac disorders) | 85 (103) | 0 (0) | 20 (24)
Pacemaker-mediated Tachycardia (PMT) (Cardiac disorders) | 0 (0) | 29 (30) | 20 (22)
Supraventricular Tachy Arrhythmia (Cardiac disorders) | 30 (34) | 29 (30) | 22 (25)
Ventricular Tachyarrhythmia (Cardiac disorders) | 26 (32) | 20 (22) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days